CLINICAL TRIAL: NCT04670263
Title: Evaluating the Efficacy of Dry Eye (DE) Disease Treatment Using Novel Tear Film Imager (TFI)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Adom Advanced Optical Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SZMC-TFI-2019
Record Dates: First submitted 2020-11-29; First posted 2020-12-17 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding will take place at the reading center: the patient measurements will be unidentified. Adom's interpreter will not know to which group the examinee belonged to. After the conclusion of the study, the blindness will be removed, and a retrospective statistical analysis will be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Eye Disease (Experimental): Subjects who will be diagnosed at baseline with Dry Eye Disease according to standard diagnosis
  Interventions: Device: Tear Film Imager
- Healthy (Active Comparator): Subjects who will be diagnosed at baseline with no Dry Eye Disease according to standard diagnosis
  Interventions: Device: Tear Film Imager

INTERVENTIONS:
Device: Tear Film Imager — Tear Film Imager recording

SUMMARY:
Dry Eye disease signs and symptoms are reduced in patients who receive topical steroids and topical hyaluronic acid.

AdOM's Tear Film Imager measurements are reproducible and it can diagnose the dry eye disease state in a single, non-invasive measurement. The Tear Film Imager can provide objective accurate measurements of the dry eye treatment effectiveness.

DETAILED DESCRIPTION:
80 subjects will be enrolled , 40 of which with positive signs and symptoms of Dry eye and 40 healthy subjects without sign and no symptoms of Dry eye. Healthy and Dry eye groups will be age- matched.

Over a period of 4 weeks, the subjects diagnosed with dry eye will be treated and as follows:

1. Hylo-comod artificial tears (0.1 % sodium hyaluronate) 8 times a day for 4 weeks
2. Coll STERODEX (Dexamethasone sodium phosphate 0.1% eye drops) 3 times a day for 2 weeks Healthy subjects will not receive any treatment.

Both groups will be examined at baseline and 4 weeks after baseline measurement.

Treatment results will be measured by both traditional methods and by Tear Film Imager.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Be at least 18 years of age at the time of enrollment of either sex or any race.
3. Best corrected visual acuity (BCVA) of 0.7 logMAR (ie, 20/100 vision) or better in each eye as measured using a Snellen chart
4. Intraocular pressure (IOP) in the range of 5 to 22 mmHg in both eyes.
5. DE subjects will be enrolled if they manifest symptoms (OSDI >=13) and signs of clinically active dry eye disease in either eye, by at least one of:

   1. Corneal fluorescein staining - at least severe in one section or moderate at two
   2. TBUT =< 10 sec
   3. Schirmer wetting of less than 10 mm in 5 min (with anesthesia).
6. Control will be enrolled if they manifest NO symptoms (OSDI <13) and NO signs of clinically active dry eye disease in either eye, by meeting all the following criteria's:

   1. Corneal fluorescein staining - negative
   2. TBUT > 10
   3. Schirmer wetting of more than 10 mm in 5 min (with anesthesia).
7. A negative urine pregnancy test if female of childbearing potential.

Exclusion Criteria:

1. Any ocular condition that could affect study parameters (glaucoma, nystagmus, keratoconus, follicular conjunctivitis, iritis or post LASIK, LASEK or PRK).
2. Have had any ocular infection within the last 30 days and/or have preauricular lymphadenopathy.
3. Any significant illness that could be expected to interfere with study parameters.
4. Use of any investigational product or device within one month prior to Visit 1 or during the study period.
5. Concomitant use of any prohibited medication (antihistamines, corticosteroids, all ocular medications or anti-allergic therapies) during the trial.
6. Any history of, positive HIV, hepatitis B, C, or evidence of acute active hepatitis A (anti HAV IgM), Any known history of iritis/uveitis, glaucoma, or other chronic ophthalmologic disorder other than allergic conjunctivitis.
7. History of any ocular surgical procedure within 3 months prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-03-08 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Tear film imager measurements with be assessed for reference values for objective tests of the disease with the Tear Film Imager | 1month
  Tear film imager meuresmend will be assessed during the study visits
Verify repeatability of Tear film imager measurement | 2 hours
  The repeatability of TFI will be evaluated by comparing the reported parameters of the two TFI measurements on first visit
Compare the clinical measurements of DES to the TFI measurements | 1month
  The correlation between the clinician's measurements of Dry Eye and the corresponding Tear film imager reported parameters of interest will used to evaluate the association between the two assessments.

SECONDARY OUTCOMES:
Changes in the lipid layer thickness | from baseline to 1 month
  Change from baseline of the lipid layer thickness as measured by the Tear film imager
Changes in the Macu-aqueous layer thickness | from baseline to 1 month
  Change from baseline of the Muco-aqueous layer thickness as measured by Tear film imager

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No